CLINICAL TRIAL: NCT01994070
Title: A Randomized Crossover Trial to Evaluate Electrical Versus Chemical Cardioversion in Patients With Acute Atrial Fibrillation
Brief Title: Chemical vs Electrical Cardioversion for Emergency Department Patients With Acute Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H12-00408
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Procainamide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrical-first (Active Comparator): Patients in atrial fibrillation for less than 48 hours will be administered procedural sedation and analgesia and an electrical current applied across their chest (cardioversion) to attempt conversion to normal sinus rhythm. If this does not succeed, they will be given intravenous procainamide (chemical cardioversion). If procainamide is required, physicians will be informed as follows: "50% of patients convert to normal sinus rhythm within one hour and 90% of patients convert within two hours." Physicians can then proceed at their discretion.
  Interventions: Drug: Electrical-first
- Chemical-first (Active Comparator): Patients in atrial fibrillation for less than 48 hours will be administered intravenous procainamide (chemical cardioversion) to attempt conversion to normal sinus rhythm. If procainamide is required, physicians will be informed as follows: "50% of patients convert to normal sinus rhythm within one hour and 90% of patients convert within two hours." Physicians can then proceed at their discretion. If this does not succeed, patients will be administered procedural sedation and analgesia and an electrical current applied across their chest (electrical cardioversion) to attempt conversion to normal sinus rhythm.
  Interventions: Drug: Chemical-first

INTERVENTIONS:
Drug: Electrical-first — Patients will be placed on cardiopulmonary blood pressure monitoring, and sedated with propofol 0.5 - 1.0 mg / kg. Once a Ramsay Sedation Scale score of 5 or greater is reached, the physician will attempt synchronized electrical cardioversion with 100 J, 200 J, 200 J. If the patient converts to normal sinus rhythm by the third shock, the physician may discharge the patient. If atrial fibrillation is maintained, the patient will receive intravenous procainamide 17 mg / kg over 30 minutes. If the rhythm has changed from atrial fibrillation to normal sinus within one hour, the attending physician may discharge the patient, otherwise a cardiologist will be consulted.
  Other Names: DC cardioversion
  Arms: Electrical-first
Drug: Chemical-first — Patients will be placed on cardiopulmonary blood pressure monitoring, and will receive intravenous procainamide 17 mg / kg over 30 minutes. If the rhythm has changed from atrial fibrillation to normal sinus within one hour, the attending physician may discharge the patient. If the rhythm has not changed, then the patient will be continue to have cardiopulmonary monitoring, but also be attended by a respiratory therapist. The patient will be sedated with propofol 0.5 - 1.0 mg / kg. Once a Ramsay Sedation Scale score of 5 or greater is reached, the physician will attempt synchronized electrical cardioversion with 100 J, 200 J, 200 J. If the patient converts to normal sinus rhythm by the third shock, the physician may discharge the patient, otherwise a cardiologist will be consulted.
  Other Names: procainamide
  Arms: Chemical-first

SUMMARY:
Atrial fibrillation (AF) is the most common type of irregular heartbeat in emergency department (ED) patients. If the irregular heartbeat has been present for less than 48 hours, there is a chance that emergency treatment can convert the heartbeat into normal rhythm.

There are currently two options for accomplishing this; both are widely and safely used in EDs. Each has its advantages and disadvantages. This study will compare the two methods. (1) Patients are given an intravenous medication called procainamide; this converts patients into a normal heart rhythm around 50% of the time. (2) Patients are sedated (put to sleep with a general anesthetic) for about ten minutes, while an electrical current is conducted across the chest; this converts patients into a normal heart rhythm around 90% of the time.

Procainamide can cause low blood pressure in about 10% of patients; this is usually corrected by administering intravenous fluids. Sedation can cause low blood pressure in about 10% of patients, and breathing trouble in about 10% of patients; this is usually corrected by administering intravenous fluids, and administering more oxygen, respectively. In thousands of patients studied around the world, there does not appear to have been a reported stroke or death as a result of these procedures.

A physician will choose one method, but if it fails, will move to the next method. There are thus two options. (1) Chemical conversion, followed by electrical conversion; and (2) Electrical cardioversion, followed by chemical cardioversion. These options both have a 90%+ chance of converting AF into a normal heart rhythm. However, the investigators believe that an electrical-chemical sequence will be faster than a chemical-electrical sequence, while both will be equally safe.

If patients agree to take part in the study, they will be randomized to one of the two options. They will have their breathing, oxygen levels, blood pressure, and heartbeat monitored for their entire ED stay.

The investigators plan to enrol 86 patients at five hospitals over the course of about one year. The primary outcome of ED length-of-stay, as well as secondary outcomes, such as conversion to normal rhythm, and adverse events (such as trouble breathing or low blood pressure) will be documented. In addition, an investigator will contact you at three and thirty days after your visit to make sure that there are no problems. Importantly, although the principal and site investigators will be aware of the primary outcome, attending emergency physicians who actually provide patient care will NOT be aware of the primary outcome--otherwise this could bias patient management.

When the study is finished, the results will be given to the writing committee merely as the "A" and "B" arms, and not specified as either the "chemical-first" or "electrical-first" arms. The writing committee will compose two manuscripts, (1) assuming that "A" is the "chemical-first" arm and "B" the "electrical-first" arm, and (2) assuming that "A" is the "electrical-first"arm, and "B" the "chemical-first" arm. After both manuscripts have been approved by all authors, the blinding will be removed and only the correct manuscript submitted for publication.

ELIGIBILITY:
Inclusion Criteria:

* Must have an abnormal heart rhythm diagnosed as AF for less than 48 hours.
* Be eligible for cardioversion (in the judgment of the study doctor).
* Are on the appropriate blood thinner medications.
* Have systolic blood pressure (SBP) above 90 mmHg and less than 160 mmHg and diastolic blood pressure (DBP) less than 95 mmHg at screening and baseline.
* Are adequately hydrated (in the judgment of the study doctor) and have a normal saline intravenous established and it is working properly.
* Must have a body weight between 45 and 136 kg inclusive (99 and 300 lbs).
* Be able and willing to give informed consent.

Exclusion Criteria:

* Pregnant or nursing a child
* Are diagnosed with any other serious lung, liver, metabolic, kidney, gastrointestinal, central nervous system, or psychiatric disease, infection, having a fever, end stage disease states, or any other diseases that could interfere with the conduct of this study. Your study doctor will confirm this with you.
* Have an infection or fever
* Are allergic to procainamide (the chemical conversion agent) or propofol (the sedative agent)
* Are participating in another drug study or have received an experimental drug within 30 days prior to screening in this study
* Are not currently living in the Vancouver Coastal Health Region
* Are unable or unwilling to be contacted at 30 days by one of the study doctors or study staff to determine 30-day outcomes
* Are unwilling to sign the informed consent form
* Are unable to speak English

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Length-of-stay | up to 12 hours
  Length of stay is defined as the time from patient randomization to discharge from the emergency department.

SECONDARY OUTCOMES:
Adverse events | up to 12 hours after randomization
  * Sentinel risk
    * Oxygen desaturation > 60 seconds or < 75%
    * Apnea > 60 seconds
    * Shock
    * Cardiac arrest
  * Minor risk
    * Oxygen desaturation < 60 seconds
    * Apnea < 20 seconds
    * Airway obstruction
    * Failed sedation
    * Allergic reaction, no anaphylaxis
    * Bradycardia
    * Tachycardia
    * Hypotension
    * Hypertension
    * Ventricular arrhythmia
    * Seizure
  * Minimal risk
    * Vomiting / retching
    * Subclinical respiratory depression
    * Muscle rigidity
    * Hypersalivation
    * Paradoxical response
    * Recovery agitation
    * Prolonged recovery
  Note: All potential adverse events will be referred to a central safety committee. Members of this committee will be blinded to patient treatment group and blinded to 3- and 30-day outcomes. The central safety committee will determine whether an adverse event occurred and categorize the severity.

OTHER OUTCOMES:
Quality of life | 30 days
  Patients will be contacted by telephone three and 30 days after the ED visit and asked quality of life questions based on the Short Form (SF)-8. The 30-day outcomes of stroke and death will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Scheuermeyer, MD, Principal Investigator — St. Paul's Hospital
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada